CLINICAL TRIAL: NCT05019612
Title: The Role of Expectations on Complaints and Well-being After Endometriosis Surgery
Brief Title: The Role of Expectations on Complaints and Well-being After Endometriosis Surgery in Women
Acronym: ROXWELL
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Helmut Schmidt University (Other)
Collaborators: Frauenklinik an der Elbe (Unknown)
Responsible Party: Principal Investigator, Dr. Yvonne Nestoriuc, Prof., Helmut Schmidt University
Other Study IDs: ROXWELL-2021-HH
Record Dates: First submitted 2021-08-16; First posted 2021-08-25 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Endometriosis; Expectations; Laparoscopy
Keywords: cohort study; endometriosis; surgery; laparoscopy; expectation; nocebo; placebo
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- single-group/one cohort: Women with endometriosis, having the clinical indication for laparoscopic endometriosis excision
  Interventions: Procedure: Laparoscopy: A minimal invasive surgery

INTERVENTIONS:
Procedure: Laparoscopy: A minimal invasive surgery — A low-risk minimal invasive surgery performed in the pelvis using small incisions. With the aid of a laparoscope, the operator views the affected area in real-time. Beyond that, the camera sends images to a video monitor. The operator obtains endometriosis and biopsy samples with small surgical instruments. Before laparoscopy, individuals are provided with a general anaesthetic to relax muscles and prevent pain during surgery.

SUMMARY:
Endometriosis is a prevalent disease in women of procreative age. Most endometriosis patients are affected in their daily life by complaints such as chronic pelvic pain, dysmenorrhoea, infertility, or pain during sexual intercourse. Yet, its etiology is poorly understood. Although laparoscopy is well known as the gold standard for treating endometriosis, 20-30% of treated women still show persistent complaints following successful laparoscopy.

It has been widely recognized that expectations profoundly affect treatment courses and outcomes in many different health conditions. Additionally, evidence suggests that optimizing preoperative expectations can improve post-operative outcomes such as disability and return to work.

The objective of this study is to investigate whether expectations also affect treatment course and outcome in women after endometriosis surgery. For this purpose, the investigators conduct a mixed-method observational cohort study to gather data on psychological factors, particularly treatment and symptom-related expectations, as well as complaints and well-being of patients after surgery. A sample of N = 300 women will be asked pre- and postoperatively to evaluate these psychological factors and indicators of treatment course and outcome. Overall, the study will last 12 months, including one assessment preoperatively (baseline), seven monthly assessments postoperatively, and a follow-up assessment 12 months after endometriosis surgery.

The study aims to determine potential interactions between aforementioned psychological factors, their influence on the postoperative health, and the long- and short-term symptom course of patients with endometriosis. The study results will provide a better understanding of the symptom- and treatment course in women with endometriosis and subsequently supply clinical approaches to optimize treatment of endometriosis.

DETAILED DESCRIPTION:
Rationale:

According to the evidence-based S2-treatment guidelines for endometriosis, laparoscopy is the method of choice to remove endometriosis and is associated with considerable symptom improvement. However, 20-30% of treated women (so-called non-responders) still report symptoms and impairments after surgery; this is not explainable by laparoscopy itself or a recurrence of endometriosis. Relevant psychosocial predictors are higher age and pain catastrophization, though both only explain a small amount of persistent symptoms and impairments. This indicates a potential role of other psychological factors influencing treatment outcome, such as expectations.

Evidence for this assumption is provided by placebo-response rates of 30% in women who had a sham endometriosis surgery and even reported symptom improvements after diagnostic (sham) laparoscopy. Concerning other gynaecological settings, research already implies that expectations have a remarkable impact on treatment outcome and quality of life in women with breast cancer. Likewise, the role of expectations could be important for the optimal treatment of endometriosis.

However, there is no study examining the role of expectations on treatment outcomes in women with endometriosis to date. Therefore, this study investigates the influence of expectations and other psychological factors on complaints and well-being of patients after surgery in women with endometriosis.

Method:

In the proposed study, a sample of 300 women will report pre- and postoperatively about their treatment and symptom expectations, health condition, and other psychological factors that may influence treatment course and outcome after endometriosis surgery. Overall, this monitoring will last 12 months, including one assessment preoperatively (baseline), seven monthly assessments postoperatively, and a follow-up assessment 12 months after endometriosis surgery. All assessments will be conducted online.

Within the scope of an embedded qualitative study, a partial sample of 20 to 30 women will be interviewed preoperatively and postoperatively about their treatment and symptom expectations, fears, and concerns regarding the laparoscopy.

Above that, a second partial sample of 20 women will report on seven consecutive days about their current health condition, and treatment and symptom expectations in their everyday life using ambulatory assessment (smartphone-based measurements).

Objectives:

Firstly, the investigators are interested in the treatment course and outcome and its possible changes over a period of six months after endometriosis surgery. Secondly, the role of pre- and post-operative expectations for treatment course and outcome for women with endometriosis should be determined. Besides expectations, the investigators will finally examine further potential psychological and social predictors for treatment outcome, e.g., prior treatment experiences, state anxiety, depression, pain catastrophization and demographics, in order to optimize endometriosis therapy.

Regarding the embedded qualitative study, the investigators explore and categorize the mentioned treatment- and symptom-related expectations concerning endometriosis surgery (laparoscopy) and psychological factors that potentially improve or harm women's treatment outcome and health condition. The ambulatory assessment offers a monitoring of patients' symptom course in their daily lives and the determination of potential modulators

ELIGIBILITY:
Inclusion Criteria:

1. Adult women (18+)
2. Endometriosis related symptoms and complaints
3. Clinical indication for surgery/laparoscopy
4. Clinically diagnosed endometriosis (postoperatively)
5. Informed consent
6. Sufficient knowledge of the German language

Exclusion Criteria:

1. Incomplete excision of endometriosis
2. Malignant biopsy result (postoperatively)

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Endometriosis is a chronic disease affecting individuals of the female biological sex
Study Population: Women will be selected who are treated in the Frauenklinik an der Elbe.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-08-25 (Actual); Primary Completion 2024-06-20 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
Course of Endometriosis related Pain Disability - Pain Disability Index (PDI-D) | at baseline, seven times consecutive with an interval of four weeks, follow-up 12 months after surgery
  The PDI-D assesses the self-reported disability by endometriosis symptoms using a numeric rating scale with eleven response options (0-10). The overall total score will be calculated by gathering all seven items. The course of endometriosis related pain disability over the measurement points will be analysed as the primary outcome.

SECONDARY OUTCOMES:
Severity of endometriosis-related complaints - self-conducted rating scale (NRScomplaints) | at baseline, seven times consecutive with an interval of 4 weeks, follow up 12 months after surgery
  The NRScomplaints Questionnaire assesses the self-reported severity of the five most prevalent endometriosis symptoms (dysmenorrhoea, pelvic pain, dyspareunia, dyschezia, dysuria) by a numeric rating scale with eleven response options (0-10). The overall total score will be examined.
Mental well-being - Short Warwick-Edinburgh Mental Wellbeing Scale (SWEMWBS) | at baseline, seven times consecutive with an interval of four weeks, follow up 12 months after surgery
  The SWEMWBS assesses the self-reported mental well-being using seven statements about thoughts and feelings with five response (1=never to 5=always) options. The total score ranges from 7 to 35, higher sum scores reflect a higher level of mental well-being.
Health related quality of life - Endometriosis Health Profile (EHP-5) | at baseline, seven times consecutive with an interval of 4 weeks, follow up 12 months after surgery
  The EHP-5 measures the wide range of effects that endometriosis can have on women's lives covering five items with five response options (0=never to 4=always). A higher sum score reflects a higher level of self-reported impairment.
Current Treatment effects - 'Generic rating scale for treatment effects' (GEEE_ACT) | Continuous measurement postoperatively, seven times with an interval of four weeks
  The GEEE_ACT assesses the self-reported current treatment effects on endometriosis related complaints using three numeric rating scales with eleven response options (0-10). The total sum score will be examined.

OTHER OUTCOMES:
Impairments by somatic symptoms - Patient Health Questionnaire (PHQ-15) | at baseline, seven times consecutive with an interval of four weeks, follow up 12 months after surgery
  The PHQ-15 assesses patients' self-reported impairment and consists of 15 physical symptoms with eleven response options (0-10). The total score ranges from 0 to 30, with higher scores indicating more impairment.
Treatment expectations - Treatment Expectation Questionnaire (TEX-Q) | at baseline
  The TEX-Q measures patients' self-reported treatment expectations and consists of 15 items with eleven response options (0-10). The total score ranges from 0 to 150 with higher scores implying more positive treatment expectations.
Expected Endometriosis Pain Disability - Pain Disability Index, adapted (PDI-expect) | at baseline, seven times consecutive with an interval of four weeks, follow up 12 months after surgery
  The PDI-expect assesses the expected disability by endometriosis symptoms using a numeric rating scale with eleven response options (0-10). The overall total score will be examined by gathering all seven items.
Symptom expectation - self-conducted rating scale (NRS_Symptomexpect) | at baseline, seven times consecutive with an interval of four weeks, follow up 12 months after surgery
  The NRSSymptomexpect Questionnaire assesses the expected symptom severity of the five most prevalent endometriosis symptoms (dysmenorrhoea, pelvic pain, dyspareunia, dyschezia, dysuria) using a numeric rating scale with eleven response options (0-10). The overall total score will be examined.
Pre-experiences with endometriosis treatment/surgery - Generic rating scale for previous treatment experiences (GEEE_PRE) | at baseline
  The GEEE_PRE is a self-reported measure to assess previous experiences with endometriosis treatment/surgery. If experience with endometriosis surgery is indicated, three items are presented to rate the experiences on a numeric analogue scale (0-10). The total sum score will be examined.
Treatment expectations - Generic rating scale for treatment expectations (GEEEEXP) | at baseline, seven times consecutive with an interval of four weeks, follow up 12 months after surgery
  The GEEE_EXP assesses treatment expectations related to endometriosis surgery using three numeric rating scales with eleven response options (0-10). The total sum score will be examined.
Depressive and anxiety - Patient Health Questionnaire (PHQ-4) | at baseline
  The PHQ-4 comprises four items, inquiring the degree to which an individual experiences anxiety or a depressed mood through a four-level likert scale (0-3). The overall total score ranges from 0 to 12. A higher sum score indicates a higher level of state anxiety and depression.
Pain Catastrophization - subscale of the Coping- strategy questionnaire (CSQ-D) | at baseline
  The Pain catastrophization subscale assesses pain catastrophization, compromising six items with seven response options (0=never do that to 6=always do that). A total score will be examined. A higher sum score indicates a higher level of pain catastrophization.

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Nestoriuc, Prof. Dr., Principal Investigator — Helmut Schmidt University/ University of the Federal Armed Forces Hamburg
Locations (1):
- Helmut Schmidt University, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in published articles will be shared after deidentification via a repository. A study protocol is available.
  Audio records will be deleted, transcripts are available following publications upon reasonable request.
Supporting Information: Study Protocol
Time Frame: Data will be available when the main research questions were answered by the investigators.
Access Criteria: Anyone who whishes to access the quantitative data. Transcripts are available upon reasonable request.

REFERENCES:
- [Background] von Blanckenburg P, Schuricht F, Albert US, Rief W, Nestoriuc Y. Optimizing expectations to prevent side effects and enhance quality of life in breast cancer patients undergoing endocrine therapy: study protocol of a randomized controlled trial. BMC Cancer. 2013 Sep 18;13:426. doi: 10.1186/1471-2407-13-426. PMID 24047450
- [Background] Heisig SR, Shedden-Mora MC, von Blanckenburg P, Schuricht F, Rief W, Albert US, Nestoriuc Y. Informing women with breast cancer about endocrine therapy: effects on knowledge and adherence. Psychooncology. 2015 Feb;24(2):130-7. doi: 10.1002/pon.3611. Epub 2014 Jun 21. PMID 24953538
- [Background] Nestoriuc Y, von Blanckenburg P, Schuricht F, Barsky AJ, Hadji P, Albert US, Rief W. Is it best to expect the worst? Influence of patients' side-effect expectations on endocrine treatment outcome in a 2-year prospective clinical cohort study. Ann Oncol. 2016 Oct;27(10):1909-15. doi: 10.1093/annonc/mdw266. Epub 2016 Aug 22. PMID 27551051
- [Background] Pan Y, Kinitz T, Stapic M, Nestoriuc Y. Minimizing Drug Adverse Events by Informing About the Nocebo Effect-An Experimental Study. Front Psychiatry. 2019 Jul 25;10:504. doi: 10.3389/fpsyt.2019.00504. eCollection 2019. PMID 31427995
- [Background] Quidde J, Pan Y, Salm M, Hendi A, Nilsson S, Oechsle K, Stein A, Nestoriuc Y. Preventing adverse events of chemotherapy by educating patients about the nocebo effect (RENNO study) - study protocol of a randomized controlled trial with gastrointestinal cancer patients. BMC Cancer. 2018 Sep 24;18(1):916. doi: 10.1186/s12885-018-4814-7. PMID 30249191
- [Background] Shedden-Mora MC, Pan Y, Heisig SR, von Blanckenburg P, Rief W, Witzel I, Albert US, Nestoriuc Y. Optimizing Expectations About Endocrine Treatment for Breast Cancer: Results of the Randomized Controlled PSY-BREAST Trial. Clin Psychol Eur. 2020 Mar 31;2(1):e2695. doi: 10.32872/cpe.v2i1.2695. eCollection 2020 Mar. PMID 36397978
- [Background] Nestoriuc Y, Kleine-Borgmann J. [Appearances are not deceptive: clinical evidence and new research approaches to open-label placebo]. Nervenarzt. 2020 Aug;91(8):708-713. doi: 10.1007/s00115-020-00953-6. German. PMID 32691079
- [Derived] Meyrose AK, Basedow LA, Hirsing N, Buchweitz O, Rief W, Nestoriuc Y. Assessment of treatment expectations in people with suspected endometriosis: A psychometric analysis. F1000Res. 2024 Sep 9;13:174. doi: 10.12688/f1000research.145377.2. eCollection 2024. PMID 39328391
- [Derived] Hirsing N, Meyrose AK, Buchweitz O, Nestoriuc Y. Do expectations determine postoperative disability in women with endometriosis? Study protocol for a clinical mixed-methods observational cohort study. BMJ Open. 2023 Jan 4;13(1):e067497. doi: 10.1136/bmjopen-2022-067497. PMID 36599637